CLINICAL TRIAL: NCT01473511
Title: Delivering Intervention for Pediatric Behaviour Problems at a Distance: a Randomized Trial of Strongest Families Ontario
Brief Title: Strongest Families Ontario (Formerly the Family Help Program)
Acronym: SF-ON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4839; MCT-91030 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2011-07-22; First posted 2011-11-17 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Oppositional Defiant Disorder; Behaviour Disorder
Keywords: Behavioural intervention; Distance intervention; Parenting intervention
MeSH Terms: conditions — Oppositional Defiant Disorder; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strongest Families Program + Usual care (Experimental): 50% randomized to receive Strongest Families intervention immediately as well as the usual care services available via the referring agency for the 22 month study period.
  Interventions: Behavioral: Strongest Families Intervention (formerly Family Help)
- Usual care (No Intervention): 50% randomized will not receive Strongest Families Intervention during the 22 month study phase, but will receive the usual care services available via the referring agency. At the end of the 22 month study period study participants will be offered the Strongest Families Intervention services.

INTERVENTIONS:
Behavioral: Strongest Families Intervention (formerly Family Help) — Distance HEALTH education intervention focussed on skill learning for parents
  Other Names: formerly the Family Help Program
  Arms: Strongest Families Program + Usual care

SUMMARY:
Strongest Families (formerly Family Help)is an evidence-based, distance health education model for families who have children with behavioural difficulties. The principal research question is "Does Strongest Families, a 12-week, home-based program of interactive readings, instructional videos, homework projects, and weekly "coaching" telephone calls out perform the care families typically experience when referred to a mental health service?". The investigators hypothesize that children randomized to Strongest Families intervention will show a significantly greater reduction in externalizing behaviour problems than those randomized to a Control (usual care). In addition, parents randomized to Family Help will report a greater improvement in parenting skills and a greater reduction in symptoms of emotional distress (i.e., feeling of anxiety, depression, and stress) than parents in the Control condition. Finally, families randomized to Family Help will use fewer mental health services than Controls.

DETAILED DESCRIPTION:
Our project is designed to help families and children with mild or moderate symptoms early, before problems become worse and more difficult to treat.

The Strongest Families Program is a distance parenting program that was developed at the Centre for Research in Family Health at the IWK Health Centre in Halifax, Nova Scotia. Most families are able to manage these problems if they are given the skills to do so. The Strongest Families "Parenting the Active Child" Distance Program is done over the telephone; families do not have to travel to a centre to receive help. This program includes a handbook, videos and weekly phone calls between the parent and non-professional'coach'. The coach provides support to families, answer questions and guide parents as they learn the skills. Strongest Families has helped hundreds of families in Nova Scotia.

ELIGIBILITY:
Inclusion Criteria:

Male or female individuals who meet all the following criteria are eligible for this trial:

* Child is aged 6 to 12 years and
* Completed and signed referral form from a participating intake site is received and
* Parent/legal guardian provides verbal, telephone consent to participate and
* Ability of participant to read and understand English (at a Grade 5 level) and
* There must be the reasonable intention that for the study duration the child will remain in the direct care of the participant and at the same address as the participant (2 years) and o Child presents with significant levels of disruptive behaviour based on the BCFPI results at the referring agent end and clinical evaluation of the corroborative study assessment measures.

Exclusion Criteria:

Participants meeting one or more of the following criteria cannot be selected:

* Child is in the care of a child protective agency or currently being investigated by a child protective agency
* Child has received any form of behavioural treatment in the past 6 months
* Child is at an imminent risk of harm to themselves or others
* In the judgment of the investigator or delegate, any condition that may interfere with effective delivery of the study protocol/intervention program (i.e., High parental DASS-21 score, complex child symptomology, families who are unmotivated or are in complete chaos)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2010-02; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Child Behaviour Checklist | Baseline, 5, 10, 16, 22 months
  Results will be analyzed as change from baseline over time

SECONDARY OUTCOMES:
Alabama Parenting questionnaire | Baseline, 5, 10, 16, 22 months
  Results will be analyzed as change from baseline over time
SCAPI (economic) | Baseline,5, 10, 16, 22
  Results will be analyzed as change from baseline over time
DASS-21 | Baseline,5, 10, 16, 22
  Results will be analyzed as change from baseline over time
Investigator designed Satisfaction measure | end of intervention
  Participant satisfaction with this psychological intervention will be measured at the end of intervention that varies between participants, but on average is about 5 months post-randomization
Investigator designed disability measure | weekly during intervention
  Results will be analyzed as change from baseline over time
Discrete Conjoint Preference survey: Investigator designed | baseline, 5, 16 months
  We will examine if discrete choice data collected at baseline predicts participation, adherence and outcome. We will also explore changes in preferences over time.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, PhD, Principal Investigator — Vice President of REsearch Services
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate summary data would be made available but not individual data.

REFERENCES:
- [Background] Lingely-Pottie P, McGrath PJ. A therapeutic alliance can exist without face-to-face contact. J Telemed Telecare. 2006;12(8):396-9. doi: 10.1258/135763306779378690. PMID 17227604
- [Background] Lingley-Pottie P, McGrath PJ. Telehealth: a child and family-friendly approach to mental health-care reform. J Telemed Telecare. 2008;14(5):225-6. doi: 10.1258/jtt.2008.008001. PMID 18632994
- [Background] Lingley-Pottie P, McGrath PJ. Distance therapeutic alliance: the participant's experience. ANS Adv Nurs Sci. 2007 Oct-Dec;30(4):353-66. doi: 10.1097/01.ANS.0000300184.94595.25. PMID 18025870
- [Background] Lingley-Pottie P, McGrath PJ. A paediatric therapeutic alliance occurs with distance intervention. J Telemed Telecare. 2008;14(5):236-40. doi: 10.1258/jtt.2008.080101. PMID 18632997
- [Background] Lingley-Pottie P, McGrath PJ. Development and initial validation of the treatment barrier index scale: a content validity study. ANS Adv Nurs Sci. 2011 Apr-Jun;34(2):151-62. doi: 10.1097/ANS.0b013e3182186cc0. PMID 21572262
- [Background] McGrath PJ, Lingley-Pottie P, Emberly DJ, Thurston C, McLean C. Integrated knowledge translation in mental health: family help as an example. J Can Acad Child Adolesc Psychiatry. 2009 Feb;18(1):30-7. PMID 19270846
- [Background] McGrath PJ, Lingley-Pottie P, Thurston C, MacLean C, Cunningham C, Waschbusch DA, Watters C, Stewart S, Bagnell A, Santor D, Chaplin W. Telephone-based mental health interventions for child disruptive behavior or anxiety disorders: randomized trials and overall analysis. J Am Acad Child Adolesc Psychiatry. 2011 Nov;50(11):1162-72. doi: 10.1016/j.jaac.2011.07.013. Epub 2011 Sep 3. PMID 22024004
- [Background] Lingley-Pottie P, Janz T, McGrath PJ, Cunningham C, MacLean C. Outcome progress letter types: parent and physician preferences for letters from pediatric mental health services. Can Fam Physician. 2011 Dec;57(12):e473-81. PMID 22170209
- [Background] Lingley-Pottie P, McGrath PJ, Andreou P. Barriers to mental health care: perceived delivery system differences. ANS Adv Nurs Sci. 2013 Jan-Mar;36(1):51-61. doi: 10.1097/ANS.0b013e31828077eb. PMID 23370500